CLINICAL TRIAL: NCT03531307
Title: Lactate Levels at Beginning of Surgery Correlates With Ki-67 Labeling Index in Brain Tumors
Brief Title: Lactate Levels Correlates With Ki-67 in Brain Tumor Surgery
Status: Completed | Type: Observational
Sponsor: Ricard Valero (Other)
Responsible Party: Sponsor-Investigator, Ricard Valero, Head of Neuroanesthesia. Associated Professor., Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Other Study IDs: Lac001Ki67
Record Dates: First submitted 2018-04-24; First posted 2018-05-21 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Brain Tumor; Anesthesia
Keywords: Lactate; Ki-67; Mitotic index; Brain tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lactate and Ki 67 levels: Neurosurgical patients between June 2017 and February 2018 for tumoral and non-tumoral craniectomy with lactate levels at the beginning of surgery and Ki-67 index in biopsies.
  Interventions: Other: Data correlation

INTERVENTIONS:
Other: Data correlation — Correlation between lactate levels and Ki-67 index

SUMMARY:
In neurosurgery, brain tumor patients show increased levels of lactate at the beginning of surgery. This has been related to malignancy. Ki-67 is a cell proliferation index used as a marker of tumor mitotic activity.

This research aims to describe the correlation between lactate levels and the Ki-67 index in patients with brain tumor.

DETAILED DESCRIPTION:
Lactate levels are used in the evaluation of perfusion status in critical care. Increases not related to a hypoperfusion state are observed in the patient with brain tumors. These increases have been related to type and tumor grade. This observation does not fully explain the variation within the same tumor grade.

Ki-67 label index is a marker of mitotic activity that can be used as proliferation index. It has been associated with histologic grade and survival rate. Provides a quantitative measure of the tumor proliferation status.

The investigators will perform a retrospective analysis of the clinical charts of patients after brain tumor resection. The study will address the relationship between baseline lactate levels and the proliferation index found in tissues biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Neurosurgical craniectomy cases
* June 2017 - February 2018
* Valid lactate information after anesthesia induction
* Ki-67 label index informed in biopsies
* Tumor type information confirmed in biopsies

Exclusion Criteria:

* Incomplete lactate or Ki-67 index information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Craniectomy cases for tumoral and non-tumoral surgery with lactate levels and biopsy information.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the correlation between Lactate levels and Ki-67 Index | Within 1 week after data acquisition
  Levels of lactate in first blood analysis after anesthesia induction and proliferation index in biopsy results

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Valero, Dr., Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Anesthesia department, Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No